CLINICAL TRIAL: NCT02998996
Title: A Phase I/II, Randomised, Placebo-controlled, Partially-blinded, Parallel-group Study to Assess the Safety, Tolerability and Immune Response Following Vaccination With Immunose™ FLU
Brief Title: Study to Assess the Safety, Tolerability and Immune Response Following Vaccination With Immunose™ FLU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eurocine Vaccines AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EURO 15-11
Record Dates: First submitted 2016-11-10; First posted 2016-12-21 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-10

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Endocine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Immunose™ FLU 1%, (Experimental): 15 µg haemagglutinin(HA)/strain and 1% Endocine™
  Interventions: Biological: 15 µg HA/strain and 1% Endocine™
- Immunose™ FLU 2%, (Experimental): 15 µg HA/strain and 2% Endocine™
  Interventions: Biological: 15 µg HA/strain and 2% Endocine™
- Influenza antigen, (Experimental): 15 µg HA/strain
  Interventions: Biological: 15 µg HA/strain
- Saline (NaCl), (Placebo Comparator): Placebo
  Interventions: Biological: Placebo, Saline
- i.m. comparator, (Active Comparator): 15 µg HA/strain
  Interventions: Biological: intramuscular comparator
- i.n. comparator (Active Comparator)
  Interventions: Biological: intranasal comparator

INTERVENTIONS:
Biological: 15 µg HA/strain and 1% Endocine™ — intranasal administration
  Arms: Immunose™ FLU 1%,
Biological: 15 µg HA/strain and 2% Endocine™ — intranasal administration
  Arms: Immunose™ FLU 2%,
Biological: 15 µg HA/strain — intranasal administration
  Arms: Influenza antigen,
Biological: intramuscular comparator — intramuscular administration
  Arms: i.m. comparator,
Biological: intranasal comparator — intranasal administration
  Arms: i.n. comparator
Biological: Placebo, Saline — intranasal administration
  Arms: Saline (NaCl),

SUMMARY:
The main purpose of the this study is to evaluate the safety and tolerability of Immunose™ FLU based on Endocine™ and quadrivalent influenza antigen.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study related procedures.
* Male or female 18-39 years of age (both inclusive) at screening
* Subjects who the Investigator believes will comply with the requirements of the protocol.
* BMI: 18.0 and 30.0 kg/m2 (inclusive).
* Judged by the Investigator to have no serious illness based on medical history, physical examination, ECG, vital signs and blood and urine assessments at screening.
* From the signing of the informed consent until 2 months after the last vaccination (Visit 3 for group 1 to 4 and Visit 2 for group 5 and 6) female subjects have to use contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen- only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD], intrauterine hormone-releasing system [IUS], bilateral tubal occlusion, sexual abstinence). Any male partner should be willing to use condom or should be vasectomized.

Exclusion Criteria:

* Diagnosis of laboratory-confirmed influenza in the 2015/2016 season.
* Use of any investigational drug product within 3 months before screening or planned use during the study period, including the safety follow-up.
* Administration of an influenza vaccine during the 6 months before screening.
* Previously received another vaccine within 28 days before administration of the study vaccine, or is scheduled to receive another vaccine during the study period, excluding the safety follow-up.
* Any contra-indication to intramuscular administration of the influenza vaccine AdimFlu-S according to its prescribing information.
* Any contra-indication to administration of the influenza vaccine Fluenz Tetra according to its summary of product characteristics (SmPC).
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to eggs or egg product as well as ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin, gentamycin and neomycin sulphate).
* Diagnosis of asthma with poor disease control as assessed by the Investigator.
* Potent immunosuppressive therapy including cytostatics, antibodies, drugs acting on immunophilins, interferons and other drugs used to prevent rejection of organ transplants, within 6 months before screening.
* Use of any parenteral or oral corticosteroids within 30 days prior to screening. Inhaled steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any progressive or severe neurologic disorder, seizure disorder or Guillain-Barré syndrome.
* History of Guillain-Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Received blood, blood products and/or plasma derivatives or any administration of immunoglobulin preparation within the three months prior to Visit 2, or planned during the study.
* Participation in blood donation within 3 months or plasma donation within 1 month prior to Visit 2.
* History of substance or alcohol abuse within the past 2 years.
* History or any illness/condition that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.
* Pregnant or lactating female or intent to become pregnant during the clinic phase (up until and including Visit 4 for group 1 to 4 and Visit 3 for group 5 and 6) and for 2 months after the last vaccination.
* History of Bell's palsy.
* Ongoing regular use of intranasal sprays including corticosteroids and decongestants.
* Ongoing cough, sinusitis, allergic rhinitis, nasal polyps or obstruction, including septum deviation significant enough to prevent bilateral administration of study vaccine.
* Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Subjects that are prone to nosebleed.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Lif-Tiberg, MD, Principal Investigator — CTC
Locations (2):
- Sweden (2):
  - Site 2, Linköping
  - Site 1, Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immunose™ FLU 1%, | Immunose™ FLU 2%, | Influenza Antigen, | Saline (NaCl), | i.m. Comparator, | i.n. Comparator
Started | 36 | 35 | 36 | 18 | 18 | 19
Completed | 36 | 34 | 35 | 18 | 17 | 19
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Family reasons | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunose™ FLU 1%, | Immunose™ FLU 2%, | Influenza Antigen, | Saline (NaCl), | i.m. Comparator, | i.n. Comparator | Total
Number analyzed (Participants) | 36 | 35 | 36 | 18 | 18 | 19 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 36 | 18 | 18 | 19 | 162
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.36 (5.69) | 26.34 (5.46) | 25.11 (4.8) | 27.72 (5.6) | 27.22 (4.75) | 24.68 (4.32) | 26.13 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 20 | 15 | 9 | 8 | 91
  Male | 16 | 16 | 16 | 3 | 9 | 11 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African descent | 0 | 2 | 0 | 1 | 0 | 0 | 3
  Ethnicity: Asian or Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Ethnicity: Caucasian | 35 | 32 | 34 | 17 | 17 | 19 | 154
  Ethnicity: Mixed/multi-racial | 0 | 1 | 2 | 0 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Sweden | 36 | 35 | 36 | 18 | 18 | 19 | 162

OUTCOME MEASURES:

1. Primary Outcome: Local Tolerability - First Dose
Description: Local tolerability, as measured by at least one of the administration site reactions swelling, redness, pain and pruritus, regardless of severity.
Time Frame: Pre-dose, and 15 and 120 min after study drug administration (Visit 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Immunose™ FLU 1%, | Immunose™ FLU 2%, | Influenza Antigen, | Saline (NaCl), | i.m. Comparator, | i.n. Comparator
Number analyzed (Participants) | 36 | 35 | 36 | 18 | 18 | 19
Participants
  Pre-dose | 5 | 4 | 9 | 0 | 0 | 4
  15 min post-dose | 11 | 10 | 7 | 0 | 9 | 3
  120 min post-dose | 9 | 5 | 7 | 0 | 6 | 1

2. Primary Outcome: Local Tolerability - Second Dose (Group 1-4 Only)
Description: as for outcome 1
Time Frame: Pre-dose, and 15 and 120 min after second study drug administration (Visit 3).
Measure: Count of Participants; unit: Participants
Arm/Group | Immunose™ FLU 1%, | Immunose™ FLU 2%, | Influenza Antigen, | Saline (NaCl),
Number analyzed (Participants) | 36 | 35 | 36 | 18
Participants
  Pre-dose | 8 | 8 | 7 | 2
  15 min post-dose | 16 | 12 | 10 | 2
  120 min post-dose | 10 | 8 | 5 | 1

ADVERSE EVENTS:
Time Frame: From first dose of IMP until the subject's last visit to the clinic (Visit 4 for Group 1 to 4 and Visit 3 for Group 5 and 6). In addition to collection of AEs at the clinic visits, solicited and unsolicited AEs were collected using a diary for 10 days after each dose administration. SAEs and AEs of special interest were also collected during 6 months after the last vaccination.
Arm/Group | Immunose™ FLU 1%, | Immunose™ FLU 2%, | Influenza Antigen, | Saline (NaCl), | i.m. Comparator, | i.n. Comparator
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35 | 0/36 | 0/18 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/36 | 0/35 | 0/36 | 0/18 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 32/36 | 30/35 | 26/36 | 10/18 | 13/18 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunose™ FLU 1%, (N=36) | Immunose™ FLU 2%, (N=35) | Influenza Antigen, (N=36) | Saline (NaCl), (N=18) | i.m. Comparator, (N=18) | i.n. Comparator (N=19)
Eryipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunose™ FLU 1%, (N=36) | Immunose™ FLU 2%, (N=35) | Influenza Antigen, (N=36) | Saline (NaCl), (N=18) | i.m. Comparator, (N=18) | i.n. Comparator (N=19)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (7) | 8 (9) | 1 (1) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (25) | 20 (31) | 13 (19) | 1 (1) | 2 (2) | 7 (9)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal muscosal disorder (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 7 (8) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (8) | 8 (14) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (28) | 13 (23) | 10 (16) | 5 (7) | 3 (3) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 10 (12) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 12 (20) | 7 (9) | 3 (3) | 3 (3) | 4 (5)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (15) | 12 (17) | 2 (4) | 2 (2) | 4 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 22 (38) | 21 (38) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 10 (18) | 10 (17) | 14 (17) | 3 (4) | 5 (5) | 6 (8)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 6 (7) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 1 (3)
Fatigue (General disorders) | 13 (22) | 13 (22) | 14 (22) | 5 (8) | 8 (8) | 4 (6)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 9 (11) | 2 (3) | 4 (6) | 1 (1) | 2 (2) | 1 (1)
Swelling (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (9) | 2 (6) | 4 (5) | 3 (4) | 2 (2) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 5 (5) | 2 (3) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 6 (7) | 1 (1) | 4 (4) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02998996/Prot_SAP_000.pdf